CLINICAL TRIAL: NCT05433753
Title: Asian Multicenter Prospective Study in HER2 Positive Early Breast Cancer for Detecting Minimal Residual Disease by Circulating Tumor DNA Analysis With Neoadjuvant Chemotherapy; HARMONY Study
Brief Title: Asian Multicenter Prospective Study in HER2 Positive Early Breast Cancer for Detecting MRD by ctDNA;HARMONY Study
Status: Recruiting | Type: Observational
Sponsor: National Cancer Center, Japan (Other Government)
Responsible Party: Sponsor
Other Study IDs: NCCH2113
Record Dates: First submitted 2022-06-07; First posted 2022-06-27 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assess minimal residual disease (MRD) in HER2-positive early breast cancer patients in Asian countries. The purpose is to evaluate the relation between the detection rate of MRD and recurrence.

DETAILED DESCRIPTION:
This study will evaluate the relation between the detection rate of minimal residual disease(MRD) and recurrence in HER2-positive early breast cancer patients in Asian countries. Blood will be regularly collected to check the presence of ctDNA in HER2-positive breast cancer patients who have scheduled for neoadjuvant chemotherapy followed by surgery. Prognostic data is also collected on the same patients.

MRD is a small number of cancer cells left in the body during or after treatment. These cells have the potential to cause recurrence in cancer patients. MRD detection can help identify patients at increased risk of disease recurrence and guide treatment decisions. However, limited data are available on when ctDNA analysis should be done in the course of treatment, and what is the appropriate analysis method. This study will contribute to determining whether MRD detection using ctDNA is useful to predict the recurrence of HER2-positive early breast cancer patients. If this can be proven, it is expected that detection of MRD can use as a biomarker to assist in the de-/escalation of treatment strategies, therefore allowing to avoid overtreatment in patients at low risk, and to add more intensive treatment in patients at high risk. Moreover, studying with Asian countries, the results will become the basic data for approval of liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20 years or older at the date of registration.
2. Histological diagnosis of HER2-positive invasive breast carcinoma.
3. Patients scheduled for neoadjuvant chemotherapy followed by surgery.
4. Clinical Stage IIA-IIIC.
5. Known hormone receptor status.
6. Signed informed consent.

Exclusion Criteria:

1. Any other malignancy within 5 years prior to registration, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the esophagus, stomach, colon, or cervix.
2. Bilateral synchronous breast cancer.
3. History of breast cancer.
4. Pregnancy at registration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive early breast cancer patients who have scheduled for neoadjuvant chemotherapy followed by surgery.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (IDFS) | The duration from the date of surgery until the date of first documented the IDFS events, whichever comes first, up to 3 years.
  ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer

SECONDARY OUTCOMES:
Overall survival (OS) | The duration from the date of surgery until the date of death from any cause, up to 3 years.
  Death attributable to any cause
Disease-free survival (DFS) | The duration from the date of surgery until the date of first documented the DFS events, whichever comes first, up to 3 years.
  IDFS events, ipsilateral or contralateral DCIS, second primary non-breast invasive cancer

CONTACTS AND LOCATIONS:
Overall Officials: Sho Shiino, MD, PhD, Principal Investigator — Department of Medical Oncology, National Cancer Cancer Hospital
Locations (1):
- National Cancer Center Hospital, Japan, Chuo-ku, Tokyo, Japan